CLINICAL TRIAL: NCT02517164
Title: Role of Vitamin D Levels (Serum 25-hydroxyvitamin D) and Cognitive Impairment in the Occurrence of Falls
Acronym: VITADCOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 11-053
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Accidental Falls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum 25-hydroxyvitamin D
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fallers: patients aged 50 years and over who already fell
  Interventions: Other: Measurement of serum 25-hydroxyvitamin D; Other: Analysis of global cognitive efficiency score assessed by the "Montreal Cognitive Assessment" (MoCA).
- At risk of falls: patients aged 50 years and over at risk of falls
  Interventions: Other: Measurement of serum 25-hydroxyvitamin D; Other: Analysis of global cognitive efficiency score assessed by the "Montreal Cognitive Assessment" (MoCA).

INTERVENTIONS:
Other: Measurement of serum 25-hydroxyvitamin D
Other: Analysis of global cognitive efficiency score assessed by the "Montreal Cognitive Assessment" (MoCA).

SUMMARY:
Every year, nearly 30% of people aged over 65 fall at least once and about 15% fall at least twice. These falls can have serious consequences that are a significant threat to the independence and well-being of older people. From an economic perspective, the cost of medical care related to falls and resulting injuries is very high and continue to grow with the aging of the population. Therefore falls prevention is a public health priority.

Many data suggest that cognitive, common disorders in the elderly, is a major risk factor for falls and the elderly often have difficulty managing their parallel postural stability and other situations requiring attentional resources. Furthermore, the data used to evoke a role of vitamin D in the risk of falls in the elderly. Indeed, vitamin D has beneficial effects on muscle and on the human brain and several recent studies have shown the existence of positive relationship between serum 25 hydroxyvitamin D and cognitive function. These different actions may explain the beneficial effect of vitamin D supplementation on the risk of falling for practicing daily oral doses of vitamin D in the range of 700-1000 IU.

Our goal in this study is to confirm the existence of a link between vitamin D status and some areas of cognitive functions, and analyze the roles played by vitamin D deficiency and cognitive impairment in the occurrence of falls. The study will also seek the existence of a threshold level of 25-hydroxyvitamin D below which may arise cognitive disorders. The prospective follow-up of patients for 2 years will study the effect of correcting the vitamin D deficiency (initial correction and regular supplementation) on cognitive function, balance, walking and the occurrence of falls.

The study will be conducted in 150 subjects aged 50 years and over and fell in 150 subjects aged 50 and over at risk of falling. These patients will be enrolled in the Emergency Services, Orthopedics, Geriatrics, and Rheumatology of the University Hospital of Caen. All subjects will receive a dose of 25 hydroxyvitamin D, a comprehensive study of cognitive function, tests of balance and walking and assessment of activities of daily living and depression. All the examinations and tests will be carried out during the same half day. According to current recommendations, it will be prescribed a treatment with Vitamin D to subjects with a lowered rate of 25 hydroxyvitamin D (<30 ng / ml) to normalize the rate and will be advised doctors to prescribe regular supplementation vitamin D in order to maintain it in the standard rate (30 to 80 ng / ml). The effect of the correction of hypovitaminosis D, confirmed by controlling the rate of 25 hydroxyvitamin D, on cognitive functions, balance and walking will be analyzed 3 months and 9 months. During the two years following their inclusion in the study, subjects will be contacted by a phone call every 3 months during which will be recorded any falls they have been victims, as well as changes to their drug treatments, particularly case of regular intake of vitamin D supplementation.

If our hypothesis were true, it would be appropriate to consider a new approach to prevention of fractures involving the correction of vitamin D deficiency, cognitive rehabilitation and cognitive-motor drive in subjects with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, aged at least 50 years;
* Patient able to walk only 15 m, possibly helped by wearing a cane;
* For those aged 50 and over and having fallen: the victim of a fall from a height of uncomplicated fracture in the last 12 months; the fall occurred while standing, or walking, or from the sitting position;
* For those aged 50 and over at risk of falling: woman aged 75 and over, or about having one or more predisposing factors for falls, such as trouble walking or balance (test score the "timed up and got" ≥ 14 sec, muscle weakness of the lower limbs (≤ 4/5), visual disturbance (scale "Monoyer"; corrected visual acuity <10/20 for the sum of the two eyes), impaired lower limb proprioception (position sense test toes), depression (justifying drug therapy), cognitive disorders (MMS ≤ 26), parkinsonism (known diagnosis and clinical examination), osteoarthritis disrupting travel (known diagnosis and clinical and radiographic examinations), subject taking more than 4 drugs per day, taking psychotropic drugs.

Exclusion Criteria:

* The subject is a person deprived of liberty or an adult placed under guardianship;
* The inclusion of the subject in another biomedical research protocol for this study (unless prior approval of the principal investigator);
* The subject can walk only with the help of a third person or with the help of two canes or a walker;
* The subject is suffering from severe or progressive neurological condition;
* The subject has severe cognitive impairment (MMS <20)
* The subject has significant visual disturbances (corrected visual acuity <6/20 for the sum of 2 eyes)
* The subject received a "loading dose" of vitamin D in the last 6 months (≥ 100,000 IU);
* For subjects who dropped:

  * The fall was caused by a third party (eg stampede);
  * The subject has not dropped its height (eg fall from a ladder);
  * At the time of the fall, the subject ran or rolled cycling;
  * The fall is the result of an accident of the public highway;
  * The fall was the cause of a fracture;
  * The last drop was more than 12 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fallers and person at risk of falls aged at least 50 years
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D | change over baseline, 3 month, 9 month
"Montreal Cognitive Assessment" (MoCA). | change over baseline, 3 month, 9 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France